CLINICAL TRIAL: NCT03489005
Title: A Randomized, Double-blind, Placebo-controlled and Open-label, Active Controlled, 4 Period Crossover Trial to Evaluate the Effect of BIA 5 1058 on Cardiac Repolarization in Healthy Adult Males and Females Under Fed Conditions
Brief Title: Effect of BIA 5 1058 on Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-51058-115; 2017-001682-25 (EudraCT Number)
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Disease; Pulmonary Arterial Hypertension; Heart Failure
Keywords: BIA 5-1058; Pulmonary arterial hypertension; Heart failure; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Arterial Hypertension; Heart Failure | interventions — zamicastat; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Period 1 (Other): Interventions to be administered:
  Schema 1:
  1. 400 mg BIA 5-1058
  2. 1200 mg BIA 5-1058
  3. Placebo
  4. Moxifloxacin
  Schema 2:
  1. 1200 mg BIA 5-1058
  2. Placebo
  3. 400 mg BIA 5-1058
  4. Moxifloxacin
  Interventions: Drug: BIA 5-1058; Drug: Placebo Oral Tablet; Drug: Moxifloxacin 400 mg
- Treatment Period 2 (Other): Interventions to be administered:
  Schema 1
  1. 1200 mg BIA 5-1058
  2. Moxifloxacin
  3. 400 mg BIA 5-1058
  4. Placebo
  Schema 2:
  1. Placebo
  2. Moxifloxacin
  3. 1200 mg BIA 5-1058
  4. 400 mg BIA 5-1058
  Interventions: Drug: BIA 5-1058; Drug: Placebo Oral Tablet; Drug: Moxifloxacin 400 mg
- Treatment Period 3 (Other): Interventions to be administered:
  Schema 1
  1. Placebo
  2. 400 mg BIA 5-1058
  3. Moxifloxacin
  4. 1200 mg BIA 5-1058
  Schema 2
  1. 400 mg BIA 5-1058
  2. 1200 mg BIA 5-1058
  3. Moxifloxacin
  4. Placebo
  Interventions: Drug: BIA 5-1058; Drug: Placebo Oral Tablet; Drug: Moxifloxacin 400 mg
- Treatment Period 4 (Other): Interventions to be administered:
  Schema 1
  1. Moxifloxacin
  2. Placebo
  3. 1200 mg BIA 5-1058
  4. 400 mg BIA 5-1058 Schema 2
  1. Moxifloxacin 2. 400 mg BIA 5-1058 3. Placebo 4. 1200 mg BIA 5-1058
  Interventions: Drug: BIA 5-1058; Drug: Placebo Oral Tablet; Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: BIA 5-1058 — Subjects will receive BIA 5-1058 tablets (containing 100 mg) as single, oral doses 30 minutes after the start of a moderate mealas follows:
  * 400 mg BIA 5 1058, as 4 × 100 mg tablets and 8 placebo tablets
  * 1200 mg BIA 5 1058, as 12 × 100 mg tablets
  Other Names: Zamicastat
Drug: Placebo Oral Tablet — Matching placebo tablets administered as follows:
  - placebo, as 12 × 0-mg tablets
Drug: Moxifloxacin 400 mg — Administered as follows:
  - 400 mg moxifloxacin, as 1 × 400-mg tablet

SUMMARY:
The purpose is to evaluate the effect of single therapeutic (400 mg) and supratherapeutic (1200 mg) doses of BIA 5-1058 on the time-matched change from baseline in placebo-adjusted interval corrected (QT) for heart rate (HR)

DETAILED DESCRIPTION:
This will be a Phase 1, randomized, double-blind, placebo-controlled and open-label, active controlled, 4 period, crossover study in healthy male and female subjects under fed conditions.

The study will be double blinded for BIA 5-1058 and placebo and open label for moxifloxacin. The central ECG laboratory and ECG readers will be blinded to study treatment sequence, timepoint, and subject. All subjects will receive each of the following 4 treatments:

* 400 mg BIA 5 1058
* 1200 mg BIA 5 1058
* placebo
* 400 mg moxifloxacin

Potential subjects will be screened to assess their eligibility to enter the study between 28 and 3 days prior to the first treatment administration. For each treatment period, subjects will be admitted into the Clinical Research Unit (CRU) on Day 2 and be confined to the CRU until Discharge on Day 4. Each subject will receive a single dose of study medication on Day 1 of each treatment period. There will be a washout of at least 10 days between doses, and subjects will return to the CRU for a Follow-up visit 14 ± 2 days after Period 4 Discharge. The total duration of study participation for each subject from Screening through Follow-up visit) is anticipated to be approximately 80 days.

The start of the study is defined as the date the first enrolled subject signs an Informed Consent Form (ICF). The point of enrollment occurs at the time of subject number allocation. The end of the study is defined as the date of the last subject's last assessment (scheduled or unscheduled).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 28.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is acceptable) at Screening or Period 1 Check-in as assessed by the Investigator (or designee).
* No clinically significant abnormalities in 12-lead ECG rate, rhythm, or conduction at Screening or Period 1 Check-in.
* Females will not be pregnant (negative pregnancy test at Screening and Period 1 Check in) or lactating, and females of childbearing potential and males will agree to use contraception.
* Able to comprehend and willing to sign an ICF before any study procedure and to abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* Increased risk if dosed with moxifloxacin, according to the product label for moxifloxacin.
* History of tendonitis or tendon rupture associated with treatment with quinolone antibiotics.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
* Subjects with alanine aminotransferase >1.0 × the upper limit of normal (ULN) and/or aspartate aminotransferase >1.0 × ULN and/or total bilirubin >1.0 × ULN (isolated bilirubin >1.0 × ULN and ≤1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%), as confirmed by subsequent repeat assessment, at Screening or Period 1 Check-in.
* Sustained supine systolic blood pressure >140 mmHg or <90 mmHg or diastolic blood pressure >95 mmHg at Screening or baseline for Period 1 unless deemed not clinically significant by the Investigator.
* A resting ECG HR <45 bpm or >90 bpm.
* An abnormal ECG indicating a second- or third-degree atrioventricular block, or one or more of the following: QRS interval >110 ms, QTcF <300 ms or >450 ms, or PR interval >220 ms. Any rhythm other than sinus rhythm that is interpreted by the Investigator to be clinically significant.
* History of additional risk factors for torsades de pointes (eg, heart failure, hypokalemia) or a family history of long QT syndrome or sudden death.
* History of clinically significant alcoholism or drug/chemical abuse.
* Alcohol consumption of >28 units per week for males and >21 units per week for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
* Positive alcohol breath test result, positive urine cotinine test, or positive urine drug screen (confirmed by repeat) at Screening or Period 1 Check-in.
* Positive hepatitis panel and/or positive human immunodeficiency virus test. Subjects whose results are compatible with prior immunization may be included at the discretion of the Investigator.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to the first dose.
* Use or intend to use any medications/products known to alter QT/QTc within 14 days or 5 half-lives (whichever is longer) prior to the first dose, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to the first dose, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any prescription medications/products including hormone replacement therapy and oral, implantable, transdermal, injectable, or intrauterine hormonal contraceptives within 14 days prior to the first dose, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any slow-release medications/products considered to still be active within 14 days prior to the first dose, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to the first dose, unless deemed acceptable by the Investigator (or designee).
* Use of tobacco- or nicotine-containing products within 3 months prior to Screening.
* Receipt of blood products within 2 months prior to Period 1 Check-in.
* Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
* Vegetarians, vegans, or other medical dietary restrictions.
* Subjects who do not have suitable veins for multiple venipunctures/cannulation as assessed by the Investigator.
* Have previously completed or withdrawn from this study or any other study investigating BIA 5 1058, and have previously received the investigational product.
* Not able to reliably communicate with the Investigator or sub-Investigator.
* Unlikely to cooperate with the requirements of the study.
* Subjects who are study site employees or immediate family members of a study site or Sponsor employee.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
time-matched change from baseline in placebo-adjusted QT interval corrected for heart rate based on an individual correction method after BIA 5-1058 dosing. | Day 1 at -1.25, -1, and -0.75 hours predose, Day -1 (baseline) at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hours and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 23 hours postdose.
  In each treatment period, continuous 12-lead digital ECG recording will be performed by Holter monitor for at least 24 hours prior to dose until approximately 24 hours postdose.

SECONDARY OUTCOMES:
QT interval corrected for heart rate based on the Fridericia correction (QTcF) | Day 1 at -1.25, -1, and -0.75 hours predose, Day -1 (baseline) at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hours and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 23 hours postdose.
  In each treatment period, continuous 12-lead digital ECG recording will be performed by Holter monitor for at least 24 hours prior to dose until approximately 24 hours postdose.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided